CLINICAL TRIAL: NCT02504164
Title: Effect of Midazolam Premedication on the Satisfaction Levels of Patients After Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2014-0310
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Early Gastric Cancer; Gastric Adenoma
Keywords: midazolam; satisfaction; endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms; Personal Satisfaction | interventions — Midazolam; Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No premedication (Experimental): No premedication before sedation
  Interventions: Drug: No premedication
- Midazolam (Active Comparator): Premedication with midazolam before sedation
  Interventions: Drug: midazolam 0.02mg/kg

INTERVENTIONS:
Drug: midazolam 0.02mg/kg
  Other Names: Premedication of midazolam 0.02mg/kg before sedation for endoscopic submucosal dissection
  Arms: Midazolam
Drug: No premedication — No premedication before sedation for endoscopic submucosal dissection
  Arms: No premedication

SUMMARY:
Endoscopic submucosal dissection is commonly performed under light to moderate sedation, and minimizing patient movement is of key importance for successful outcome. Propofol has widely replaced benzodiazepines as sedative drug of choice, and has been reported to enhance the quality of procedure in our past study. However, despite higher satisfaction scores of the endoscopists and faster post-procedural recovery, patient satisfaction scores were found to be higher in patients that received midazolam and meperidine instead of propofol and remifentanil. This seems to be due to the anterograde amnestic effects of midazolam rather than the quality of sedation itself. Investigator hypothesized that by premedicating the patient with low lose midazolam before receiving sedation for ESD with propofol and fentanyl, patient satisfaction would be enhanced without affecting endoscopic performance.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over the age of 19 diagnosed with early gastric cancer or gastric adenoma that are scheduled for endoscopic submucosal dissection
2. American society of anesthesiologist physical status 1~3

Exclusion Criteria:

1. Patient refusal
2. Patients that received sedatives within 24 hours prior to endoscopic submucosal dissection
3. History of gastrectomy or previous endoscopic submucosal dissection at same site
4. Allergies to propofol or its ingredients, soybeans or peanuts
5. Pregnant or breastfeeding patients
6. Patients with severe debilitating underlying medical conditions
7. Patients with altered mental status
8. Illiterate patients or foreigners

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction scores on a scale from 0 to 10 | 24 hours after ESD
Willingness to receive same method of sedation for ESD in the future as yes or no | 24 hours after ESD
Post-procedural pain on a VAS scale of 0 to 10 | at 1 hour and 24 hours after ESD
Any recall of the ESD procedure on a scale from 0 to 2 (0; no recall, 1; partial recall, 2; can recall most of procedure) | 24 hours after ESD

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea